CLINICAL TRIAL: NCT07303595
Title: Effect of a Postpartum Multivitamin-Mineral Supplement on Maternal Nutrient Status and Wellbeing
Brief Title: Mom Multi Postnatal Supplementation Trial
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Perelel Inc. (Industry)
Collaborators: University of Georgia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: PROJECT00012011; Sponsor (Other: Perelel Health)
Record Dates: First submitted 2025-09-02; First posted 2025-12-26 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-12

CONDITIONS: Postnatal Care
Keywords: Postnatal; multivitamin dietary supplement

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Multivitamin supplement pack (Experimental): 4 capsules and 1 softgel
  Interventions: Dietary Supplement: Perelel Mom Multi
- Placebo (Placebo Comparator): 4 capsules + 1 softgel
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Perelel Mom Multi — Daily Perelel postnatal multivitamin supplement throughout intervention
  Arms: Multivitamin supplement pack
Dietary Supplement: Placebo — Daily placebo capsules throughout intervention
  Arms: Placebo

SUMMARY:
The goal of this clinical trial is to learn if a vitamin and mineral supplement designed specifically for women after childbirth can improve their nutrition and health in women who are pregnant or have recently given birth (within 6 weeks).

The main question it aims to answer is:

Can a postpartum-specific vitamin and mineral supplement help improve nutritional status and health outcomes in women after giving birth?

Researchers will compare women who take the new postpartum vitamin and mineral supplement to women who take a placebo (fake pills without active ingredients) to see if the supplement improves their nutritional health.

Participants will:

Attend 2 visits at University of Georgia (1-1.5 hours each) over 12 weeks Participate in 2 phone calls between visits Stop taking other vitamin/mineral supplements during the study Have blood drawn to test vitamin and mineral levels Provide urine samples and breastmilk samples if breastfeeding (optional) Have height, weight, and skin color measured Complete questionnaires about health, pregnancy, and mental wellness Answer questions about daily food and drink intake Take either the study supplement or placebo daily

ELIGIBILITY:
Inclusion criteria:

* Healthy, postpartum women (~4 weeks [± 2 weeks]) with infants born term and singleton
* Not pregnant during the study period
* Able to understand (written and spoken) English or Spanish.

Exclusion criteria:

* Cardiometabolic disease
* Past pregnancy complications (gestational diabetes, hypertension)
* malabsorption syndromes (IBS, IBD, Crohn's, Colitis, Celiac)
* Caily use of medications which may affect nutrient absorption
* chronic alcohol use (> 4 alcoholic drinks/day)
* those prescribed postnatal MVM supplements by their physician
* unwilling to discontinue dietary supplementation containing any of the active components in the study product over the study period
* Women should not have an allergy or intolerance to active or inactive product ingredients.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-11-10 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
To assess the effects of the multi-vitamin-mineral (MVM) supplement on changes in maternal Vitamin D status as compared to placebo among healthy, postpartum women. | 12 weeks
  Changes in serum Vitamin D (25-hydroxyvitamin D (25(OH)D) from baseline to end of intervention (12 weeks)
To assess the effects of the multi-vitamin-mineral (MVM) supplement on changes in maternal iron status as compared to placebo among healthy, postpartum women. | 12 weeks
  Changes in Iron status (serum iron, ferritin, TIBC, transferrin) from baseline to end of intervention (12 weeks)
To assess the effects of the multi-vitamin-mineral (MVM) supplement on changes in maternal Vitamin B12 status as compared to placebo among healthy, postpartum women. | 12 weeks
  Changes in serum B12 from baseline to end of intervention (12 weeks)
To assess the effects of the multi-vitamin-mineral (MVM) supplement on changes in maternal iodine status as compared to placebo among healthy, postpartum women. | 12 weeks
  Iodine status measured as Maternal Urinary Iodine Concentrations + Creatinine at baseline and 12 weeks
To assess the effects of the multi-vitamin-mineral (MVM) supplement on changes in maternal Omega-3 status as compared to placebo among healthy, postpartum women. | 12 weeks
  Changes in RBC Omega-3 (Total, DHA, and EPA) from baseline to end of intervention (12 weeks)
To assess the effects of the multi-vitamin-mineral (MVM) supplement on changes in maternal folate status as compared to placebo among healthy, postpartum women. | 12 weeks
  Changes in folate status (RBC folate) from baseline to end of intervention (12 weeks)

SECONDARY OUTCOMES:
To assess the effects of the MVM supplement on changes in maternal mental health/wellbeing questionnaire among healthy, postpartum women. | 12 weeks
  Change in scores on WHOQOL-BREF questionnaire of maternal mental health/wellbeing outcomes from baseline to end of 12 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- UGA Clinical & Translational Unit, Athens, Georgia, United States